CLINICAL TRIAL: NCT01071980
Title: Work Place Adjusted Intelligent Physical Exercise Reducing Musculoskeletal Pain in Shoulder and Neck (VIMS) - Industrial Workers
Acronym: VIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: University of Copenhagen (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Lars L. Andersen, Senior Researcher, PhD, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: VIMS00
Record Dates: First submitted 2010-01-25; First posted 2010-02-19 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Non-specific Pain of the Neck and Shoulder

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Specific resistance training (Active Comparator): 3 x 20 min a week of specific resistance training for 20 weeks
  Interventions: Other: Work Place Adjusted Intelligent Physical Exercise Reducing Musculoskeletal Pain in Shoulder and Neck
- Control (No Intervention): Control group

INTERVENTIONS:
Other: Work Place Adjusted Intelligent Physical Exercise Reducing Musculoskeletal Pain in Shoulder and Neck — Participants will be randomized at the cluster level to a control group or 20 weeks of specific resistance training for 3 x 20 min a week
  Arms: Specific resistance training

SUMMARY:
The purpose of this study is to investigate the effect of specific resistance training on neck/shoulder pain in industrial workers.

ELIGIBILITY:
Inclusion Criteria:

* industrial worker

Exclusion Criteria:

* trauma, life threatening diseases, pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Pain of the neck and shoulders | At week 0 (baseline) and week 20 (follow-up)
Pain in the arm/hand | At week 0 (baseline) and week 20 (follow-up)

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Centre for the Working Environment, Copenhagen, Denmark

REFERENCES:
- [Derived] Pedersen MT, Andersen CH, Zebis MK, Sjogaard G, Andersen LL. Implementation of specific strength training among industrial laboratory technicians: long-term effects on back, neck and upper extremity pain. BMC Musculoskelet Disord. 2013 Oct 9;14:287. doi: 10.1186/1471-2474-14-287. PMID 24106771
- [Derived] Andersen CH, Andersen LL, Pedersen MT, Mortensen P, Karstad K, Mortensen OS, Zebis MK, Sjogaard G. Dose-response of strengthening exercise for treatment of severe neck pain in women. J Strength Cond Res. 2013 Dec;27(12):3322-8. doi: 10.1519/JSC.0b013e31828f12c6. PMID 23478473
- [Derived] Roessler KK, Rugulies R, Bilberg R, Andersen LL, Zebis MK, Sjogaard G. Does work-site physical activity improve self-reported psychosocial workplace factors and job satisfaction? A randomized controlled intervention study. Int Arch Occup Environ Health. 2013 Nov;86(8):861-4. doi: 10.1007/s00420-012-0823-z. Epub 2012 Oct 14. PMID 23064844
- [Derived] Pedersen MM, Zebis MK, Langberg H, Poulsen OM, Mortensen OS, Jensen JN, Sjogaard G, Bredahl T, Andersen LL. Influence of self-efficacy on compliance to workplace exercise. Int J Behav Med. 2013 Sep;20(3):365-70. doi: 10.1007/s12529-012-9239-0. PMID 22622819
- [Derived] Andersen LL, Jakobsen MD, Pedersen MT, Mortensen OS, Sjogaard G, Zebis MK. Effect of specific resistance training on forearm pain and work disability in industrial technicians: cluster randomised controlled trial. BMJ Open. 2012 Feb 13;2(1):e000412. doi: 10.1136/bmjopen-2011-000412. Print 2012. PMID 22331386
- [Derived] Zebis MK, Andersen LL, Pedersen MT, Mortensen P, Andersen CH, Pedersen MM, Boysen M, Roessler KK, Hannerz H, Mortensen OS, Sjogaard G. Implementation of neck/shoulder exercises for pain relief among industrial workers: a randomized controlled trial. BMC Musculoskelet Disord. 2011 Sep 21;12:205. doi: 10.1186/1471-2474-12-205. PMID 21936939